CLINICAL TRIAL: NCT03912766
Title: Serum Copeptin as a Predictor of the Risk of Hyponatremia After Transurethral Prostatectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Other Study IDs: MULodz 2/2016
Record Dates: First submitted 2019-04-05; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: transurethral prostatectomy; copeptin; hyponatremia; risk prediction
MeSH Terms: conditions — Prostatic Hyperplasia; Diabetes Insipidus; Hyponatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma for lab assessements required by the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transurethral Prostatectomy: male patients undergoing transurethral prostatectomy (TURP) for benign prostatic hyperplasia, routine surgical removal using resectoscope
  Interventions: Diagnostic Test: serum copeptin

INTERVENTIONS:
Diagnostic Test: serum copeptin — routine surgical method using resectoscope inserted into the urinary bladder

SUMMARY:
Hyponatremic hypovolemia is a frequent complication of transurethral resection of the prostate gland (TURP). Copeptin has been established as is a surrogate marker of vasopressin and is measured useful for thea clinical assessment of various sodium and water disturbances. The aim of our the study was to assess the utility of serum concentration of copeptin (CPP) and brain natriuretic peptide (NT-proBNP) for the prediction of postoperative alterations of serum sodium concentration. Study population comprised 43 patients with benign prostatic hyperplasia (BPH) undergoing transurethral resection of the prostate gland. In a forward stepwise multiple regression only serum copeptin before the surgery and the duration of TURP significantly explained the variation of sodium concentration for 12 hours from the start of the surgery. Serum NT-proBNP before the surgery did not predict hyponatremia 12 hours after TURP.Conclusion Serum copeptin before TURP surgery but not NT-proBNP may be a clinically useful marker of a decrease of serum sodium after TURP surgery.

DETAILED DESCRIPTION:
Introduction.Hyponatremic hypovolemia is a frequent complication of transurethral resection of the prostate gland (TURP). Copeptin has been established as is a surrogate marker of vasopressin and is measured useful for thea clinical assessment of various sodium and water disturbances. The aim of our the study was to assess the utility of serum concentration of copeptin (CPP) and brain natriuretic peptide (NT-proBNP) for the prediction of postoperative alterations of serum sodium concentration.

Methods. Study population comprised 43 patients with benign prostatic hyperplasia (BPH) undergoing transurethral resection of the prostate gland (TURP) Serum sodium and copeptin (CPP) were measured before the procedure and 12 hours after its completion. and sSerum NT-proBNP was assessment at baseline. Total amount of fluids and sodium administered intravenously and to flush the bladder during TURP was calculated in each patient. Receiver operator characteristics (ROC) curve analysis was used to determine the value of of copeptin (CPP) and NT-proBNP for that could prediction of the decrease of serum sodium after TURP

ELIGIBILITY:
Inclusion Criteria:

- glomerular filtration rate estimated from serum creatinine with CKD-EPI formula (eGFR) >45 ml/min.

Exclusion Criteria:

* acute infection
* heart failure (NYHA stage 3 or 4)
* diabetes insipidus
* nephrogenic diabetes insipidus
* other sodium homeostasis abnormalities
* impaired consciousness
* psychogenic polydipsia
* alcohol abuse.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male patients with benign prostatic hyperplasia (BPH) who wre undergoing transurethral resection of the prostate (TURP)
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
change of serum sodium after surgery | change of serum sodium from baseline to 12 hours post surgery
  predictive value of serum copeptin measured before surgery for serum sodium change after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michal Nowicki, MD PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Nephrology, Hypertension and Kidney Transplantation, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided
whole dataset could be shared if required and justified by research interest